CLINICAL TRIAL: NCT05895448
Title: Treatment of Recent Injection Drug Use With Chronic HCV Infection in U.S. Liver Referral Clinics: A Prospective, Observational Cohort Study And Contemporaneous Therapy Cohort Without Injection Drug Use
Brief Title: Treatment of HCV-Infected Recent Injection Drug Users in U.S. Liver Clinics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center For Hepatitis C, Atlanta, GA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1364-2018
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Chronic Hepatitis C; People Who Inject Drugs
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — velpatasvir

STUDY DESIGN:
Intervention Model Description: PWID arm and non-PWID arm prospective, parallel observational cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PWID (people who inject drugs) (Experimental): velpatasvir (100 mg) and sofosbuvir (400 mg) once daily for 12 weeks (brand or branded generic) in subjects who had used intravenous drugs at least once in preceding six months.
  Interventions: Drug: velpatasvir and sofosbuvir once daily for 12 weeks (brand or branded generic) .
- Non-PWID (Active Comparator): velpatasvir (100 mg) and sofosbuvir (400 mg) once daily for 12 weeks (brand or branded generic) in subjects who had NOT used intravenous drugs at least once in preceding six months, but were treated concurrently in the same hepatology referral clinics.
  Interventions: Drug: velpatasvir and sofosbuvir once daily for 12 weeks (brand or branded generic) .

INTERVENTIONS:
Drug: velpatasvir and sofosbuvir once daily for 12 weeks (brand or branded generic) . — Directly active antiviral therapy (velpatasvir 100 mg+sofobuvir 400 mg) once daily

SUMMARY:
Direct antiviral therapy (standard of care) administered to chronic hepatitis C-infected patients, in two hepatology clinics, who had used intravenous drugs in the past 6 months of signing informed consent (IC). This cohort was compared to concurrently treated chronic hepatitis C patients who were not intravenous drug users, who signed IC in these same clinics. Follow-up expected two years after cure and relapse rates recorded.

Primary end point was SVR rate and secondary end points included reinfection rates in follow-up period.

DETAILED DESCRIPTION:
Chronically HCV-infected participants were recruited and treated at two liver referral clinics in Georgia, but had been referred from opioid substitution therapy clinics, primary care and GI clinics, neighboring hospitals, and correctional centers. Once consented, a nurse navigator was assigned to each participant was responsible for all subjects' appointments, and med supplies. Drug testing was mandated at specified intervals. Patients with recent injection drug use (within 6 months) were assigned to the PWID (people who inject drugs) arm, and those who hadn't injected within 6 months, but agreed to be in the study and signed consents, were assigned to the non-PWID arm. Both groups were treated with velpatasvir (100 mg) and sofosbuvir (400 mg) once daily for 12 weeks (brand or branded generic). Adherence was assessed by pill counts. Mandatory treatment visits were scheduled for baseline, 4 and 12 weeks (+/- 2 weeks) and follow-up (FU) week 12 (+ 4 months). Long-term FU was flexible and could be virtual, but was mandated once yearly with HCV RNA testing.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection and PWID arm: use of intravenous drug use at least once in preceding six months. In Non-PWID arm: no use of intravenous drug use at least once in preceding six months.

Exclusion Criteria:

* Co-infection with chronic hepatitis B; Decompensated cirrhosis current or by history; inability to sign informed consent; unwilling to take therapy or unable to obtain therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Response | 24 weeks after medication initiation
  Undetectable HCV RNA 12 weeks after completion of antiviral therapy

SECONDARY OUTCOMES:
Reinfection rate hepatitis C | in follow-up period (expected 2-3 years)
  Detection of HCV RNA in follow-up period after SVR has been obtained
Intravenous drug use | informed consent through end of follow-up (up to 3 years)
  rate of IV drug use compared between baseline and end of follow-up
Opioid Substitution Therapy (OST) | informed consent through end of follow-up (up to 3 years)
  rate of OST compared between baseline and end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: brian pearlman, MD, Principal Investigator — Wellstar Internal Medicine Associates
Locations (1):
- Wellstar Atlanta Medical Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No